CLINICAL TRIAL: NCT01271322
Title: Sequential FDG-PET (Positron Emission Tomography) and Induction Chemotherapy in Locally Advanced Adenocarcinoma of the Esophagogastric Junction (AEG): The Heidelberg Imaging Program in Cancer of the Oesophago-gastric Junction During Neoadjuvant Treatment: HICON Trial
Brief Title: Sequential FDG-PET (Positron Emission Tomography) and Induction Chemotherapy in Locally Advanced Adenocarcinoma of the Esophagogastric Junction (AEG)
Acronym: HICON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT200811021017
Record Dates: First submitted 2010-12-17; First posted 2011-01-06 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Adenocarcinomas of the Esophagogastric Junction
Keywords: PET; response evaluation; neoadjuvant; radiochemotherapy; adenocarcinoma of the esophagogastric junction; esophageal carcinoma; evaluation of preoperative (radio)-chemotherapy in patients with adenocarcinomas of the oesophagogastric junction
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: neoadjuvant radiochemotherapy in metabolic non responders — Metabolic non-responders, with a SUV decrease of less than 35%, discontinue induction chemotherapy and proceed to an intensified radiochemotherapy treatment

SUMMARY:
Prospective, single-center, nonrandomized, explorative imaging study evaluating the value of PET as a predictor of histopathological response in metabolic non-responders Patients with resectable AEG (adenocarcinoma of the esophagogastric junction) type I and II (cT3/4 and/or cN+ and cM0)

Metabolic non-responders, showing a <35% decrease of SUV (standardized uptake value) two weeks after the start of neoadjuvant chemotherapy are eligible for the study and are taken to intensified taxane-based RCT (radiochemotherapy) before surgery. 18FDG-PET scans will be performed before (=Baseline) and after 14 days of standard neoadjuvant therapy as well after the first cycle of Taxotere/Cisplatin chemotherapy (=PET1) and at the end of intensified radiochemotherapy (PET2).

Tracer uptake will be assessed semiquantitatively using standardized uptake values (SUV). The percentage difference Delta SUV=100(SUVBaseline-SUVPET1)/ SUVBaseline will be calculated and assessed as an early predictor of histopathological response. In a secondary analysis, the association between the difference SUVPET1 - SUVPET2 and histopathological response will be evaluated.

DETAILED DESCRIPTION:
The HICON trial is a prospective, single-center, nonrandomized, explorative imaging study evaluating the value of PET (Positron emission tomography) as a predictor of histopathological response in metabolic non-responders Patients with resectable AEG (adenocarcinoma of the esophagogastric junction) type I and II, staged cT3/4 and/or cN+ and cM0 by endoscopic ultrasound, spiral CT or MRI and FDG-PET are eligible. Tumors must be potentially R0 resectable and must have a sufficient FDG-baseline uptake. Only metabolic non-responders, showing a <35% decrease of SUV (standardized uptake value) two weeks after the start of neoadjuvant chemotherapy are eligible for the study and are taken to intensified taxane-based RCT (chemoradiotherapy (45 Gy) before surgery. 18FDG-PET scans will be performed before (=Baseline) and after 14 days of standard neoadjuvant therapy as well after the first cycle of Taxotere/Cisplatin chemotherapy (=PET1) and at the end of intensified radiochemotherapy (PET2). Tracer uptake will be assessed semiquantitatively using standardized uptake values (SUV). The percentage difference Delta SUV=100(SUVBaseline-SUVPET1)/ SUVBaseline will be calculated and assessed as an early predictor of histopathological response. In a secondary analysis, the association between the difference SUVPET1 - SUVPET2 and histopathological response will be evaluated..

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven adenocarcinoma of the distal oesophagus (AEG type I) or cardia (AEG type II) with or without metastases in local lymph nodes (tumor stage cT3/T4, cNX, and cM0 in the tumor-node-metastasis classification)
* Staging procedures include endoscopy, endoscopic ultrasound and computed tomography (CT) of the chest and abdomen.
* Eligible patients have to be fit for platin-containing chemotherapy
* Tumors must be potentially R0 resectable tumors during consecutive operation.
* Tumors must have demonstrated a minimal amount of FDG-uptake in the baseline PET-CT, defined as 18FDG-uptake in tumor at first examination > 1,35 x hepatic-SUV + 2 x standard-deviation of hepatic-SUV, and must be a metabolic non-responder under EOX, defined as a decrease of the SUVmax of <35% in a second PET on day 14 of chemotherapy.

Exclusion Criteria:

* Eastern Cooperative Oncology Group score >1
* Previous or secondary malignancy
* Life expectancy of less than 3 months
* Uncontrolled bleeding from the tumor
* Tumor infiltration of the airways
* Pregnancy
* Uncontrolled diabetes
* Patients are also ineligible if they have undergone previous chemotherapy, radiotherapy, or endoscopic laser therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Correlation between change in tumor metabolism (detected by PET) and histopathological response | PET Baseline, PET1 (before RCHT, week 5/6), histological examination of the resected tumor
  The primary objective of the study is to evaluate the change in metabolic response - as measured by the relative difference delta SUV=100(SUVBaseline-SUVPET1)/ SUVBaseline in 18F-FDG uptake after 1 cycle of intensified taxan-based chemotherapy (PET1) - relative to the 18F-FDG uptake at the baseline examination, as a predictor of histopathological response in metabolic non-responders (assessed by PET 14 days after the start of neoadjuvant therapy).

SECONDARY OUTCOMES:
distribution of change in tumor metabolism during the treatment in histological responders and non-responders | PET Baseline, PET1 (week 5/6), histological examination of the resected tumor
  investigation of the distribution of change in tumor metabolism measured with PET Baseline and PET1(∆SUV = 100 (SUVBaseline - SUVPET1) / SUVBaseline) during the treatment in histological responders and non-responders according to the Becker Score (Histomorphology and grading of regression)
accuracy of the binary prediction rule reduction in the tumor metabolism >65% vs. <65% in histopathological responders vs. non-responders | Baseline, PET1 (week 5/6), histological examination of the resected tumor
  accuracy of the binary prediction rule delta SUV >65% vs. <65% (reduction in the tumor metabolism >65% vs. <65 % between PET Baseline and PET1 in correlation with the histopathological regression accoring to the Becker Score
association between change in tumor metabolism before/after radiochemotherapy and histopathological response | PET1 (week 5/6), PET2 (before resection), histological examination of the resected tumor
  association between tumor metabolism before/after radiochemotherapy (∆SUV = 100 (SUVPET1 - SUVPET2) / SUVPET1) and histopathological response according to the Becker Score (histomorphology and grading of regression)
association between change in tumor metabolism between PET Baseline and PET1 and overall survival as well as disease-free survival | Baseline, PET1 (week 5/6), Follow Up (q3 months during the first post-operative year, q6 months during the 2nd/3rd postoperative year)
  association between change in tumor metabolism between PET Baseline and PET 1 (∆SUV = 100 (SUVBaseline - SUVPET1) / SUVBaseline)and overall survival as well as disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Lorenzen, MD, Principal Investigator — Dep. Of Medical Oncoloy, National Center for Tumor Diseases
Locations (1):
- Nationales Centrum für Tumorerkrankungen, Heidelberg, Germany

REFERENCES:
- [Derived] Lorenzen S, von Gall C, Stange A, Haag GM, Weitz J, Haberkorn U, Lordick F, Weichert W, Abel U, Debus J, Jager D, Munter MW. Sequential FDG-PET and induction chemotherapy in locally advanced adenocarcinoma of the Oesophago-gastric junction (AEG): the Heidelberg Imaging program in Cancer of the oesophago-gastric junction during Neoadjuvant treatment: HICON trial. BMC Cancer. 2011 Jun 24;11:266. doi: 10.1186/1471-2407-11-266. PMID 21702914